CLINICAL TRIAL: NCT01469936
Title: Study of the Effect of the Food Supplement PERMEAPROTECT on the Quality of Life of Patients With Fibromyalgia (a Pilot, Double-blind, Randomized, Placebo-controlled Study)
Brief Title: Effect of PERMEAPROTECT on the Quality of Life of Patients With Fibromyalgia
Acronym: L2009-03
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2010-A00971-38
Record Dates: First submitted 2011-10-28; First posted 2011-11-10 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Irritable Bowel Syndrome
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PERMEAPROTECT (Experimental)
  Interventions: Dietary Supplement: PERMEAPROTECT
- PLACEBO (Placebo Comparator)
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: PERMEAPROTECT — Composition : glutamine, curcuma, zinc, chitosan, beta carotene, Green Tea polyphenols, thiamine and folic acid.
  Duration : 5 weeks +/- 1 week.
  Dosage :
  * First Week of intervention : 1/2 stick per day
  * Second to 5th Week : 1 stick per day
  Arms: PERMEAPROTECT
Dietary Supplement: PLACEBO — Duration : 5 weeks +/- 1 week.
  Dosage:
  * First Week : 1/2 stick per day
  * Second to 5th Week : 1 stick per day
  Arms: PLACEBO

SUMMARY:
Fibromyalgia is a medical disorder characterized by chronic widespread pain, and a heightened and painful response to pressure. Fibromyalgia symptoms are not restricted to pain, leading to the use of the alternative term fibromyalgia syndrome for the condition. Other symptoms include functional gastrointestinal pain and discomfort.

The origin of these symptoms is not yet known, and a few hypotheses have been stated. One of the supposed mechanisms that may lead to gastrointestinal hypersensitivity is a chronic, low-grade, intestinal inflammation due to an increased intestinal permeability.

In this study, we hypothesise that the food supplement PERMEAPROTECT (that contains, amongst other nutrients, glutamine and curcumin) contributes to reducing the intestinal permeability and low-grade inflammation, thus improving gastrointestinal quality of life.

DETAILED DESCRIPTION:
Patients diagnosed with fibromyalgia will enter the study and follow a run-in phase during which they will all be supplemented with prebiotics, probiotics and grape fruit seed extract for 5 weeks :

* Patients that do not present a satisfactory relief of gastrointestinal symptoms (patient subjective evaluation) will enter the randomised phase after 2 weeks +/- 1 week, at day D0.
* Patients that do present a satisfactory relief of gastrointestinal symptoms (patient subjective evaluation) will exit the study at that point, and follow their usual medical care.

Patients that enter the randomised phase will be supplemented with either PERMEAPROTECT or a PLACEBO, for 5 weeks +/- 1 week. Patients will then follow a 2 weeks +/- 1 week of wash-out, during which no supplementation will be made.

Measures of the outcomes will be made :

* at Day 0 (beginning of supplementation).
* at Day 35 (+/- 7) (end of supplementation).
* at Day 49 (+/- 7) (end of follow-up, end of study)

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30 kg/m²
* Diagnosed fibromyalgia, according to the American College of Rheumatology criteria
* Functional bowel discomfort or pain
* Pre-menopausal woman with active contraception or post-menopausal woman

Exclusion Criteria:

* Allergy to one (or more) component(s) of verum or placebo.
* Disease or disease treatment that could interfere with the efficacy evaluation.
* Treatment with statin (or HMG-CoA reductase inhibitors) associated with adverse effect
* Treatment with Coumadin (or any other Vitamin K antagonists)
* Severe depression (Beck Depression Inventory score > 16)
* Recent (during the previous month) change(s) in probiotic intake (including fermented milk, kefir, ...)
* History of major gastrointestinal surgery or inflammatory bowel disease
* Pregnant, breastfeeding or intention of pregnancy in the next three month

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of the Gastrointestinal Quality of Life Index (GIQLI) at the end of the supplementation period (5 weeks), compared with baseline. | Day D0; Day D35 (+/-7)
  The Gastrointestinal Quality of Life Index is a validated questionnaire of 36 questions related to gastrointestinal pain and discomfort, including accelerated or stalled transit, assessing the impact of these symptoms on the quality of life.

SECONDARY OUTCOMES:
Improvement of the Gastrointestinal Quality of Life Index (GIQLI) at end of follow-up (2 weeks), compared with baseline | Day D0; Day D49 (+/-7)
  The Gastrointestinal Quality of Life Index is a validated questionnaire of 36 questions related to gastrointestinal pain and discomfort, including accelerated or stalled transit, assessing the impact of these symptoms on the quality of life.
Improvement of the Impact of Fibromyalgia on the Quality of life, measured by the Fibromyalgia Impact Questionnaire (FIQ), at the end of the supplementation period (5 weeks), and at end of follow-up (2 weeks), compared with baseline. | Day D0; Day D35 (+/-7); Day D49 (+/-7)
  The FIQ is a validated questionnaire measuring the specific impact of Fibromyalgia on the quality of life.
Improvement of the subjective evaluation, by the patient, of the intensity of gastrointestinal symptoms, at the end of the supplementation period (5 weeks), and at end of follow-up (2 weeks), compared with baseline. | Day D0; Day D35 (+/-7); Day D49 (+/-7)
  Measured on a 100mm scale
Improvement of the subjective evaluation, by the patient, of the satisfactory relief of gastrointestinal symptoms, at the end of the supplementation period (5 weeks), and at end of follow-up (2 weeks), compared with baseline. | Day D0; Day D35 (+/-7); Day D49 (+/-7)
  Measured by a binary response (yes/no)
Improvement of the subjective evaluation, by the patient, of the satisfactory relief of gastrointestinal pain, at the end of the supplementation period (5 weeks), and at end of follow-up (2 weeks), compared with baseline. | Day D0; Day D35 (+/-7); Day D49 (+/-7)
  Measured by a binary response (yes/no)
Reduction of the serum C-reactive Protein (usCRP), measured by the ultra-sensitive method, at the end of the supplementation period (5 weeks), and at end of follow-up (2 weeks), compared with baseline. | Day D0; Day D35 (+/-7);
Reduction of the intestinal permeability, measured by the urinary ratio of lactulose/mannitol, at the end of the supplementation period (5 weeks), and at end of follow-up (2 weeks), compared with baseline. | Day D0; Day D35 (+/-7)
  The intestinal permeability is measured by the ratio of lactulose/mannitol. A solution of lactulose and mannitol is absorbed by the patient. Total urines are collected during the next 5 hours. Urinary lactulose and mannitol concentrations are determined and the ratio calculated.
Reduction of blood oxidative stress markers (reduced glutathione, oxidized glutathione and malondialdehyde), at the end of the supplementation period (5 weeks), and at end of follow-up (2 weeks), compared with baseline. | Day D0; Day D35 (+/-7)
Improvement of the general Quality of Life, measured by the Medical Outcome Study Short Form (MOS SF-36), at the end of the supplementation period (5 weeks), and at the en of follow-up (2 weeks), compared with baseline | Day D0; Day D35 (+/-7); Day D49 (+/-7)
  Validated questionnaire measuring the impact of health status on the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Cozon, MD, Principal Investigator — Hospice Civils de Lyon, Lyon, France; Catherine Goujon, MD, Study Director — Hospices Civiles de Lyon, Lyon, France
Locations (1):
- Unité de Recherche Clinique en Immunologie de Lyon Sud, Pierre-Bénite, France